CLINICAL TRIAL: NCT02589704
Title: A Prospective, Cross Sectional Study to Evaluate the Etiology and Nutritional Status of Cerebral Palsy Patients in Turkey
Brief Title: Nutritional Status of Cerebral Palsy Patients in Turkey
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA10
Record Dates: First submitted 2015-10-19; First posted 2015-10-28 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single visit, non-interventional, cross sectional study about risk factors, etiology, nutritional status and feeding methods in CP patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than/equal to 12 months and less than 19 years of age.
* Subject is diagnosed with cerebral palsy (CP) by a physician.

Exclusion Criteria:

* Subject presents with genopathies, cardiopathies, hypothyroidism or any pathology not related to CP.
* Subject is diagnosed with CP of postnatal origin.
* Subject has other concomitant diagnoses.

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of patients at pediatric neurology outpatient clinic diagnosed with CP, 12 months to less than 19 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1123 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
prevalence of malnutrition | at enrollment
  physician assessment

SECONDARY OUTCOMES:
etiology of CP | at enrollment
  physician assessment/medical record
correlation between type of CP and nutritional status | at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Aysugul Alptekin, MD, Study Chair — Abbott Nutrition Turkey
Locations (18):
- Turkey (Türkiye) (18):
  - Adana Numune Training and Research Hospital, Adana
  - Ankara Child Health and Diseases, Hematology, Oncology Training and Research Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Gulhane Military Medical Academy, Ankara
  - Sami Ulus Maternity and Child Health and Diseases Training and Research Hospital, Ankara
  - Fırat University Medical Faculty, Elâzığ
  - Osmangazi University Medical Faculty, Eskişehir
  - Marmara Universty Pendik Training and Research Hospital, Istanbul
  - Zeynep Kamil Woman and Child Diseases Training and Research Hospital, Istanbul
  - Dr. Behçet Uz Children's Hospital, Izmir
  - İzmir Tepecik Training and Research Hospital, Izmir
  - Kahramanmaraş Sütçü İmam University Medical Faculty, Kahramanmaraş
  - Erciyes University Medical Faculty, Kayseri
  - Selçuk University Medical Faculty, Konya
  - İnönü Universty Medical Faculty, Malatya
  - Mersin University Medical Faculty, Mersin
  - Harran University Medical Faculty, Sanliurfa
  - Karadeniz Technical University Medical Faculty, Trabzon